CLINICAL TRIAL: NCT05870709
Title: ReaL wOrld, pharmaCy-assessed Adherence to New onseT Entresto® (Sacubitril/Valsartan) in Patients With Chronic Heart Failure - a Prospective Cohort Study (LOCATE-HF)
Brief Title: Real World, Pharmacy-assessed Adherence to New Onset Entresto® (Sacubitril/Valsartan) in Patients With Chronic Heart Failure
Acronym: LOCATE-HF
Status: Withdrawn | Type: Observational
Why Stopped: Terminated due to business decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BDE05
Record Dates: First submitted 2023-04-27; First posted 2023-05-23 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
Keywords: Heart failure; NIS; Germany; sacubitril; valsartan
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- sacubitril/valsartan: patient with a first ambulatory sacubitril/valsartan prescription
  Interventions: Other: sacubitril/valsartan

INTERVENTIONS:
Other: sacubitril/valsartan — There is no treatment allocation. Patients with a first ambulatory sacubitril/valsartan prescription who are interested in study participation will be enrolled.

SUMMARY:
This is a multicenter, non-interventional, single arm cohort study with prospective collection of primary data via pharmacists in community pharmacies to describe adherence to sacubitril/valsartan in study patients at the end of the study. Eligible patients with newly prescribed sacubitril/valsartan will be observed in pharmaceutical routine.

DETAILED DESCRIPTION:
The study duration will last up to about 30 weeks per patient and will consist of a approximately three visits - Baseline visit (V1), week 1-12 (V2) and week 13-30 (V3).

No exact date for visit 2 and visit 3 will be enforced, to avoid interference with usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first ambulatory sacubitril/valsartan prescription at screening
2. Internet enabled device / smartphone (patient or affiliate)
3. ≥ 18 years of age
4. Written informed consent to participate in the study

Exclusion Criteria:

1. Depression-related medication, depression-related comorbidities (patient-reported)
2. Patients with unstable acute complications or with an advanced illness likely to interfere with participation in this trial as judged by the enrolling pharmacist
3. Simultaneous participation in any interventional trial or simultaneous participation in another Novartis-sponsored non-interventional study with sacubitril/valsartan

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure who pick up their first ambulatory sacubitril/valsartan prescription in approximately 50 participating pharmacies all over Germany.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who report a MARS-5 Score of ≥ 80% related to sacubitril/valsartan at the end of the study | Visit 3, up to 30 weeks
  Percentage of patients who report a MARS-5 Score of ≥ 80% related to sacubitril/valsartan at the end of the study will be collected.
  The MARS-5 questionnaire consists of five questions measuring non-adherence ranging from "never" (5 points) to "always" (1 points), therefore the score has a range from 5 - 25 points. This score will be transformed to a percentage score so that a patient with 5 points ("always" for all answers) scores 100% whereas a patient with 25 points ("never" for all answers) scores 0%.

SECONDARY OUTCOMES:
Number of patients with pre-defined comorbidities | Baseline
  Number of patients with pre-defined comorbidities will be collected
Number of patients with worsening of HF and reason for event. | Up to 30 weeks
  Number of patients with worsening of HF and reason for event will be collected
Number of deaths | Up to 30 weeks
  Number of deaths will be collected
Number of patients by HF-treatment | Baseline
  Number of patients by HF-treatment (ACEi, ARBs, β-blockers, MRAs, diuretics, SGLT2i) will be collected
Number of patients by reason for initiation of sacubitril/valsartan | Baseline
  Number of patients by reason for initiation of sacubitril/valsartan will be collected
Number of all medications and products that the patient is currently taking on a regular basis | Baseline
  number of all medications and products that the patient is currently taking on a regular basis (including HF medication) will be collected
Change from baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline, up to 30 weeks
  It covers physical function, clinical symptoms, social function, self-efficacy and knowledge, each with different Likert scaling wording, including limitations, frequency, bother, change in condition, understanding, levels of enjoyment and satisfaction. The score ranges from 0-100, higher scores mean a better outcome
Change from baseline in weekly patient activity and quality of life (PA & QoL) questionnaire | Up to 30 weeks
  It consists of seven questions addressing physical activity and the ability to attend patient's normal life (hobbies, house work, appointments etc) within the last week.
  Physical activity is documented as time [min] / day of physical activity and time of doing sports [h] /week. Ability of attending normal life is ranged in five categories (I fully agree / I agree / neutral / I don't agree / I don't agree at all).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No